CLINICAL TRIAL: NCT01877044
Title: The Effects of Long-term Arabinoxylan Administration on Intestinal Barrier Function and Innate Immunity
Brief Title: Long-term Effects of Arabinoxylans on Intestinal Barrier Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Bouke Salden, Coordinating Investigator, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 123050
Record Dates: First submitted 2013-06-05; First posted 2013-06-13 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Obesity; Overweight
Keywords: Prebiotics; Intestinal permeability; Gut barrier function; Immunity
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo
- NAXUS 7.5 grams (Experimental): Arabinoxylan
  Interventions: Dietary Supplement: NAXUS
- NAXUS 15.0 grams (Experimental): Arabinoxylan
  Interventions: Dietary Supplement: NAXUS

INTERVENTIONS:
Dietary Supplement: NAXUS
  Arms: NAXUS 15.0 grams; NAXUS 7.5 grams
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The higher prevalence of overweight and obesity among the population contributes to increased incidences of chronic metabolic diseases. Obesity is considered a low-grade systemic inflammatory condition through 1) production of pro-inflammatory cytokines by adipose tissue and 2) alterations in intestinal microbiota composition and associated increase in intestinal permeability. Healthcare costs related to these diseases are rising; prevention or delay of onset of disorders associated with overweight is needed. Administration of wheat arabinoxylans (NAXUS), a non-digestible carbohydrate, may change the intestinal microbiota composition and have beneficial effects on gut epithelial barrier, especially on permeability and innate immune function.

Objective: To assess the effects of NAXUS on intestinal barrier function, immune system performance and metabolic control. Prebiotic properties of NAXUS will be studied. Tolerance of the product in different doses will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Overweight men/women (BMI 28-35 kg/m2)
* Besides overweight, healthy human beings
* Fasting glucose <7.0 mmol/L
* Normal HbA1c (4.4 to 6.2%)
* Consistently stable body weight for at least 6 months (± 2 kg)

Exclusion Criteria:

* Type 2 diabetes mellitus (defined as fasting plasma glucose ≥ 7.0 mmol/L);
* Gastroenterological diseases or abdominal surgery;
* Cardiovascular diseases, cancer, liver or kidney malfunction, disease with a life expectancy shorter than 5 years;
* Abuse of products; alcohol (>20 alcoholic consumptions per week) and drugs
* Smoking
* Plans to lose weight or following a hypocaloric diet;
* Use of any medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to testing;
* Regular use of laxation products;
* Use of antibiotics in the 90 days prior to the start of study.
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Known pregnancy, lactation (checked by a pregnancy test before start of study)
* Blood donation within 3 months before study period
* Prohibited use of pro-, pre- or synbiotics during study period and three months prior to start of study. A list with forbidden products will be provided (E4 PreProbiotics).
* Self-admitted HIV-positive state
* History of any side effects towards intake of pro- or prebiotic supplements of any kind

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the change from baseline intestinal barrier function at 6 weeks, by performing a gut sugar permeability test. | Baseline and after 6 weeks of administration

SECONDARY OUTCOMES:
To assess the change from baseline intestinal barrier function at 6 weeks, by assessing the tight junction structure and proteins in colonic biopsies. | Baseline and after 6 weeks of administration
  Assessment will take place by immunofluorescent labelling and Polymerase Chain Reaction quantification of zonulin-1, claudin-3, occluding, myosin light chain kinase and phosphorylated myosin light chain.
To assess the change from baseline local and systemic immune system performance at 6 weeks. | Baseline and after 6 weeks administration
  Secondary outcome will be measured by the expression of immune parameters in colonic biopsies, by multiplex cytokine analysis in blood and Peripheral Blood Mononuclear Cell stimulation assays.
To assess the change from baseline prebiotic properties at 3 and 6 weeks, by collecting faecal samples, intestinal contents and mucosal contents. | Baseline, after 3 and after 6 weeks of administration
  The microbial community composition, Short-chain Fatty Acid profiles in intestinal content and faeces and proteolytic activity markers in intestinal content and faeces will be determined.
To assess the change from baseline glucose and lipid metabolism at 3 and 6 weeks | Baseline, after 3 and after 6 weeks of adminstration
  By determining glucose, insulin and triglyceride in blood samples. Cholesterol and free fatty acids will be measured as part of general blood profiling. Moreover effects on insulin sensitivity will be estimated by measuring HOMA-IR. Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin or C-peptide concentrations.
To assess the effect of different doses of NAXUS administration on tolerance and digestive (dys)comfort. | At baseline, after 1 wk of administration, after 2 wks of administration, after 3 wks of administration, after 4 wks of administration, after 5 wks of administration, after 6 wks of administration (in total 7 times)
  Via questionnaires stool frequency, stool consistency and gastrointestinal symptoms will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: A.A.M. Masclee, Professor, Principal Investigator — Department of Internal Medicine, Division of Gastroenterology-Hepatology
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Salden BN, Troost FJ, Wilms E, Truchado P, Vilchez-Vargas R, Pieper DH, Jauregui R, Marzorati M, van de Wiele T, Possemiers S, Masclee AA. Reinforcement of intestinal epithelial barrier by arabinoxylans in overweight and obese subjects: A randomized controlled trial: Arabinoxylans in gut barrier. Clin Nutr. 2018 Apr;37(2):471-480. doi: 10.1016/j.clnu.2017.01.024. Epub 2017 Feb 3. PMID 28214040